CLINICAL TRIAL: NCT02639000
Title: Effects of Blastocyst Stage Embryo Transfer Compared With Cleavage Stage Embryo Transfer in Women ≤ 38 Years
Brief Title: Effects of Blastocyst Stage Compared With Cleavage Stage Embryo Transfer in Women Below 39 Years
Acronym: BlastoTrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 736
Record Dates: First submitted 2015-12-15; First posted 2015-12-23 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blastocyst (Experimental): Embryo transfer of at maximum 2 embryos at blastocyst stage
  Interventions: Procedure: Embryo transfer
- Cleavage (Active Comparator): Embryo transfer of at maximum 2 embryos at cleavage stage
  Interventions: Procedure: Embryo transfer

INTERVENTIONS:
Procedure: Embryo transfer — Embryo transfer of maximum of 2 embryos at cleavage or blastocyst stage

SUMMARY:
Single center randomized study including 388 women aged less than 39 years, performing in vitro fertilization, to determine if blastocyst stage (Day 5 to 6) embryo transfer (ETs) improves implantation and pregnancy rate compared with cleavage stage (Day 2 to 3) ETs.

DETAILED DESCRIPTION:
Embryos from in vitro fertilization are routinely transferred into the woman's uterus at cleavage stage (Day 2 to 3) or at blastocyst stage (Day 5 to 6).

The rational of blastocyst stage transfer is that blastocyst stage is the most biologically correct stage for embryos to be in the uterus, and longer culture in the laboratory may give the possibility to reduce the number of genetically abnormal embryos.

The investigators design a single center randomized trial, including 388 women aged less than 39 years, performing in vitro fertilization, to confront blastocyst stage embryo transfers (ETs) and cleavage stage ETs. Each patient is randomized with a non blind randomization, based on a computer model, on the first day after fertilization.

The primary outcomes are implantation and pregnancy rate. The secondary outcome is to verify if blastocyst embryo transfer leads to a higher multiple-pregnancy rate.

An interim analysis takes place at one third of the population. Follow up is of 4 weeks for implantation rate, and covers 8 weeks regarding pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* female patients undergoing IVF procedures
* age less than 39 years

Exclusion Criteria:

* less than 4 fertilized eggs in day 1 after IVF

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 388 (Actual)
Dates: Start 2010-07; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 8 weeks after inclusion
  Number of patients achieving a clinical pregnancy divided for embryo transfers

SECONDARY OUTCOMES:
Multiple pregnancy rate | 8 weeks after inclusion
  Number of multiple pregnancies divided for pregnant patients
Implantation rate | 4 weeks after inclusion
  Number of gestational sacs divided for number of transferred embryos

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Emanuele Levi-Setti, MD, Study Director — Humanitas Research Hospital Department of Gynecology, Division of Gynecology and Reproductive Medicine Humanitas Fertility Center
Locations (1):
- Paolo Emanuele Levi Setti, Rozzano (Milan), Italy

REFERENCES:
- [Background] Glujovsky D, Blake D, Farquhar C, Bardach A. Cleavage stage versus blastocyst stage embryo transfer in assisted reproductive technology. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD002118. doi: 10.1002/14651858.CD002118.pub4. PMID 22786480
- [Derived] Levi-Setti PE, Cirillo F, Smeraldi A, Morenghi E, Mulazzani GEG, Albani E. No advantage of fresh blastocyst versus cleavage stage embryo transfer in women under the age of 39: a randomized controlled study. J Assist Reprod Genet. 2018 Mar;35(3):457-465. doi: 10.1007/s10815-017-1092-2. Epub 2017 Nov 22. PMID 29168022